CLINICAL TRIAL: NCT00236444
Title: Risperidone in the Prevention of Relapse: a Randomized, Double-blind, Placebo-controlled Trial in Children and Adolescents With Conduct and Other Disruptive Behavior Disorders.
Brief Title: A Study of the Efficacy and Safety of Risperidone in the Prevention of Relapse in Children and Adolescents With Conduct and Other Disruptive Behavior Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002020
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders
Keywords: Child; adolescent; disruptive behavior disorders; risperidone; antipsychotropic agents
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to assess the efficacy and safety of risperidone as maintenance therapy to prevent symptoms of relapse in children and adolescents with conduct and other disruptive behavior disorders, who initially responded well to treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind study to compare an oral formulation of risperidone with placebo when taken daily over 24 weeks by children and adolescents with conduct and other disruptive behavior disorders. Patients who do not respond to treatment after an initial 6-week open-label phase, or do not show continued response after 12 weeks, must leave the trial and will not enter into the 24-week double-blind phase. The principal measure of efficacy is the time to symptom relapse. Relapse is assessed by changes in following measures: the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF), a measure of symptoms of conduct and other disruptive behavior disorders and Clinical Global Impression-Severity of Illness (CGI-Severity), and a measure of overall severity of illness. Efficacy assessment also includes Clinical Global Impression-Change (CGI-C), an assessment of improvement, and Visual Analogue Scale for the most troublesome symptom (VAS-MS), which is a scale ranging from not troublesome to extremely troublesome, and Children's Global Assessment Scale (C-GAS), which is an assessment of overall functioning. Safety evaluations include incidence of adverse events, physical examinations, laboratory tests (biochemistry, hematology, and urinalysis), and electrocardiograms (ECGs). The study hypothesis is that daily treatment with an oral formulation of risperidone, compared with placebo, will result in a clinically significant difference in time to relapse, and is well tolerated by children and adolescents with conduct and other disruptive behavior disorders. Oral risperidone solution (1milligram[mg]/milliliter [ml]), daily for 36 weeks. Patients weighing at least 50 kilograms start at 0.5 ml/day and may increase up to.1.5 ml/day. Patients under 50kg start at 0.25ml/day and may increase to 0.75ml/day (maximum).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet criteria of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DMS IV) for Conduct Disorder, Oppositional Defiant Disorder, or Disruptive Behavior Disorder Not Otherwise Specified
* Have a score >=24 on the Conduct Problem subscale of the Nisonger Child Behavior Rating Form (N-CBRF)
* Have no other significant and untreated or unstable medical illness such as diabetes or hypertension, no serious illness of the liver, kidney, or significant disturbances of the cardiac, pulmonary, gastrointestinal, endocrine, or neurological system.

Exclusion Criteria:

* Patients who meet the DSM-IV criteria for: Pervasive Developmental Disorder
* schizophrenia or other psychotic disorders
* Tourette's Disorder
* Generalized Anxiety Disorder
* Major Depression
* Moderate or severe mental retardation
* Substance Dependence
* Patients with a history of neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* Hypersensitivity or intolerance to risperidone
* Pregnant or nursing females, or those lacking adequate contraception

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2001-12; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Time from start of double-blind phase to relapse, using N-CBRF and CGI assessments.

SECONDARY OUTCOMES:
Comparison of ratings for risperidone and placebo on N-CBRF, CGI, and VAS-MS throughout study. Ratings on C-GAS once during each study phase. Comparison of safety profiles of risperidone and placebo (for example, adverse events, clinical and lab tests).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the efficacy and safety of risperidone in the treatment of children and adolescents with conduct and other disruptive behavior disorders — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=449&filename=CR002020_CSR.pdf